CLINICAL TRIAL: NCT04584320
Title: Qualitative and Quantitative Identification of Clostridium Butyricum and Clostridium Neonatal in the Digestive Microbiota of Premature Infants Before 34 Weeks and Developing or Not Ulcerative Necrotizing Enterocolitis (NEC) During Their Hospitalization in Neonatology
Brief Title: Identification of Clostridium Butyricum and Clostridium Neonatal in the Digestive Microbiota of Premature Infants Before 34 Weeks and Developing or Not Ulcerative Necrotizing Enterocolitis (NEC) During Hospitalization
Acronym: ECUN-2
Status: Active, not recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: NIMAO/2019-01/MdM01
Record Dates: First submitted 2020-10-01; First posted 2020-10-12 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Necrotizing Enterocolitis
Keywords: low-birth weight infant; Clostridium butyricum; Clostridium neonatale
MeSH Terms: conditions — Enterocolitis, Necrotizing

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Stool samples taken daily from nappies
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Premature neonates with necrotizing enterocolitis
  Interventions: Other: Stool sample
- Premature neonates without necrotizing enterocolitis
  Interventions: Other: Stool sample

INTERVENTIONS:
Other: Stool sample — Stools samples taken daily to test for present of Clostridium butyricum and Clostridium neonatale

SUMMARY:
The study investigators hypothesize that Clostridium butyricum and Clostridium neonatal will be more frequently found in the stool of preterm infants with ulcerative necrotizing enterocolitis compared to healthy matched control infants. Systematic daily samples should show that the kinetics of colonization precedes the onset of the pathology. Finally, the systematic ecological survey at the time of infection could help understand the mode of acquisition and transmission of these bacteria.

ELIGIBILITY:
Inclusion Criteria:

* Premature newborn with a term of birth ≤ 34 weeks of gestation admitted to the neonatology department at the CHU of Nîmes.
* Affiliated or beneficiary of a health insurance plan.
* Newborn whose parents received informed information about the study and did not express their opposition to their child's participation in the study.

Exclusion Criteria:

* Newborn with malformative digestive pathology
* Newborn baby participating in another category 1 trial

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population consists of all newborns born less than 34 weeks of gestation admitted to the neonatology department of the CHU de Nîmes.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2021-10-18 (Actual); Primary Completion 2024-11-09 (Actual); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Presence of C. butyricum | Each day of hospitalization (maximum 120 days)
  PCR
Presence of C. neonatale | Each day of hospitalization (maximum 120 days)
  PCR
Culture of C. butyricum | Each day of hospitalization (maximum 120 days)
  Growth on selective media
Culture of C. neonatale | Each day of hospitalization (maximum 120 days)
  Growth on selective media

SECONDARY OUTCOMES:
Localisation within the hospital | During hospitalization (maximum 120 days)
  Bed numbers occupied

OTHER OUTCOMES:
Age of mother | Day 0
  Years
Body mass index of mother | Day 0
  Kg/m2
Parity of mother | Day 0
Gravidity of mother | Day 0
Professional activity of mother | Day 0
  Yes/no; description
Smoking status of mother | Day 0
  Yes/no
Chronic pathology of mother | Day 0
  Yes/no, description
Allergy of mother | Day 0
  Yes/no, description
Number of years of schooling of mother | Day 0
Exposure to magnesium sulfate during pregnancy | Day 0
  Yes/no
Cause of prematurity | Day 0
Method of delivery | Day 0
  Vagina/Caesarean
Anesthesia during delivery | Day 0
  General/spinal
Mode of delivery of vaginal birth | Day 0
  Spontaneous/instrumental
Spontaneous rupture of membranes | Day 0
  Yes/no
Time of rupture of membranes before birth | Day 0
  <12h/>12h
Pathology during pregnancy | Day 0
  Yes/No; description
Birth term | Day 0
  Weeks and days
Birth weight | Day 0
  grams
Birth weight percentile | Day 0
  percentile
Birth height | Day 0
  cm
Birth height ; percentile | Day 0
  percentile
Intubation | Day 0
  Yes/no
umbilical venous catheter | Day 0
  Yes/no; duration
Epicutaneo-cava catheter | Day 0
  Yes/no; duration
Daily lipid intake per os per kilp | During hospitlization (maximum 120 days)
  g/kg
Presence of sequelae | During hospitalization (maximum 120 days)
  Yes/no
Type of sequelae | During hospitalization (maximum 120 days)
  description
Hemodynamically significant patent ductus arteriosus | During hospitalization (maximum 120 days)
  Yes/no
Type of milk | During hospitalization (maximum 120 days)
  pasteurized/fresh/artificial
Duration of milk intake | During hospitalization (maximum 120 days)
  Days
Probiotic intake duration | During hospitalization (maximum 120 days)
  Days
Types of probiotic taken | During hospitalization (maximum 120 days)
  Type
Type of antibiotics taken in post-natal period | During hospitalization (maximum 120 days)
  Type
Duration of antibiotic treatment in post-natal period | During hospitalization (maximum 120 days)
  Days
Type of vasoactive amines taken | During hospitalization (maximum 120 days)
  Type
Duration of vasoactive amine treatment | During hospitalization (maximum 120 days)
  Days
Type of any postnatal surgery | During hospitalization (maximum 120 days)
  Type
Total duration of parenteral feeding | During hospitalization (maximum 120 days)
  Days
Ibuprofen | During hospitalization (maximum 120 days)
  Yes/no
Hemodynamic shock | During hospitalization (maximum 120 days)
  Yes/no
Labile Blood Product transfusion | During hospitalization (maximum 120 days)
  Amount
antenatal corticosteroid therapy | Day 0
  Complete/incomplete
Type of post-natal corticosteroid therapy | During hospitalization (maximum 120 days)
  Type
Duration of post-natal corticosteroid therapy | During hospitalization (maximum 120 days)
  Days
Exposure to ante- and post-natal antibiotics | During hospitalization (maximum 120 days)
  Description
umbilical arterial catheter | Day 0
  Duration
Nosocomial infection | During hospitalization (maximum 120 days)
  Proven/suspected
Nosocomial infection infective agent | During hospitalization (maximum 120 days)
  name
Rectal bleeding | During hospitalization (maximum 120 days)
  Number
metabolic acidosis | During hospitalization (maximum 120 days)
  Yes/no
Volume of alimentation per kilo | During hospitalization (maximum 120 days)
Daily carbohydrate intake per os per kilp | During hospitalization (maximum 120 days)
  g/kg
Daily proteins intake per os per kilp | During hospitalization (maximum 120 days)
  g/kg
Volume of daily total alimentation | During hospitalization (maximum 120 days)
Cranial circumference | Day 0
  cm; percentile
Cranial circumference percentile | Day 0
  percentile
Other catheter | Day 0
  Type
Duration of other catheter | Day 0
  Days
Enriched maternal milk | During hospitalization (maximum 120 days)
  Maximum percentage
Milk thickening | During hospitalization (maximum 120 days)
  Duration
Chorioamnionitis | During hospitalization (maximum 120 days)
  Proven/suspected
Materno-fetal infection | Day 0
  Proven/suspected
Materno-fetal infection infective agent | Day 0
  name
pneumatosis-pneumoportia | During hospitalization (maximum 120 days)
  Yes/no
Transfer | During hospitalization (maximum 120 days)
  Yes/no
Time of occurence of ulcerative necrotizing enterocolitis | During hospitalization (maximum 120 days)
  weeks post-natal
Warning signs of ulcerative necrotizing enterocolitis | During hospitalization (maximum 120 days)
Duration of bowel rest following necrotizing enterocolitis | During hospitalization (maximum 120 days)
Bell staging of ulcerative necrotizing enterocolitis | During hospitalization (maximum 120 days)
  from IA (suspected necrotizing enterocolitis) to IIIB (advanced necrotizing enterocolitis)

CONTACTS AND LOCATIONS:
Overall Officials: Massimo De Maio, Principal Investigator — CHU Nimes
Locations (1):
- CHU de Nimes, Nîmes, France